CLINICAL TRIAL: NCT02970630
Title: Envarsus® Tablets Administered Once Daily in Combination With Everolimus in Elderly De-novo Kidney Transplant Recipients: Open-label, Multicentre, Single-arm, Pharmacokinetic and Clinical Study
Brief Title: Envarsus® Once Daily With Everolimus in Elderly Kidney Transplant Recipients: Pharmacokinetic and Clinical Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Collaborators: Cromsource (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DFIDM-1501; 2015-005640-34 (EudraCT Number)
Record Dates: First submitted 2016-10-28; First posted 2016-11-22 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Kidney Transplantation
Keywords: prophylaxis
MeSH Terms: interventions — Tacrolimus; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (1):
- Envarsus once a day, everolimus b.i.d. (Experimental): Tacrolimus tablets at starting dose of 0.07 mg/kg/day will be administered once daily in the morning.
  Everolimus tablets at starting dose of 2 mg/day (1 mg b.i.d.) will be administered twice daily, every 12 hours.
  Interventions: Drug: Tacrolimus; Drug: Everolimus

INTERVENTIONS:
Drug: Tacrolimus — once a day
  Other Names: Envarsus
Drug: Everolimus — twice daily
  Other Names: Certican

SUMMARY:
Prospective, single-arm, open-label, multicentre study with the principal aim to estimate tacrolimus pharmacokinetic parameters in elderly de-novo kidney transplant recipients of ECD (Extended Criteria Donor) kidney grafts treated with Envarsus® prolonged release tablets in combination with everolimus tablets.

ELIGIBILITY:
Inclusion Criteria:

1. Subject's written informed consent obtained prior to transplant intervention and prior to any study-related procedures;
2. Caucasian male or female subjects aged 60 or older who are receiving a primary or secondary single or dual renal transplant from a blood group compatible deceased donor;
3. Patients who are planned to receive a renal allograft by Extended Criteria Donor (ECD);
4. Patients capable of understanding the purposes and risks of the study, who can give written informed consent and who are willing to participate in and comply with the study;
5. Patients with low to standard immunological risk, who had a PRA (Panel Reactive Antibody) ≤ 20% (PRA testing according to centre's practice);
6. Body Mass Index (BMI) between 15 and 35 kg/m2 extremes inclusive;
7. Women must be postmenopausal (physiologic menopause defined as "12 consecutive months of amenorrhea") or permanently sterilized (e.g. tubal occlusion, hysterectomy or bilateral salpingectomy) to be enrolled in the study.

Exclusion Criteria:

1. Recipients of any transplanted organ other than a single or dual kidney;
2. Patients unable or unwilling to provide informed consent;
3. Male subjects with females partner of childbearing potential UNLESS they or their partner are willing to use a reliable method of contraception (see below for details) from the time of first dose administration and until 8 weeks after the last dose of study drugs. Male subjects with partners of non-childbearing potential are not required to use contraception.

   Reliable methods of contraception for male subjects and their partner of childbearing potential must be one of the following:
   1. Placement of an intrauterine device or intrauterine system
   2. Hormonal contraception (implantable, patch, oral)
   3. Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical vaults/caps) with spermicidal foam/gel/film/cream/suppository.
   4. Male sterilization (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate "True abstinence" is acceptable only if it is in line with the preferred and usual lifestyle of the subject.
4. Recipients of a bone marrow or stem cell transplant;
5. Recipients of a kidney from a cardiac death donor;
6. Recipients of a kidney from an ABO (0, A and blood cell types) incompatible donor;
7. Recipients having pre-transplant donor specific anti-HLA (Human leukocyte antigen antibodies) (DSA) or who lost the first kidney transplant because of acute rejection;
8. Recipients of a kidney with an anticipated cold ischemia time ≥ 24 hours;
9. Recipients positive for Hepatitis C virus (HCV-RNA positive) and/or Hepatitis B Virus (HBV-DNA or HBsAg positive);
10. Recipients positive for Human Immunodeficiency Virus (HIV-Ab positive);
11. Patients with a current malignancy or a history of malignancy (within the past 5 years), except basal or non-metastatic squamous cell carcinoma of the skin that has been treated successfully;
12. Patients with uncontrolled concomitant infection, a systemic infection requiring treatment, or any other unstable medical condition that could interfere with the study objectives;
13. Patients with severe diarrhoea, vomiting, active peptic ulcer or gastrointestinal disorder that may affect the absorption of study drugs;
14. Patients with a white blood cell count ≤ 2.8x109/L unless the absolute neutrophil count (ANC) is ≥ 1.0x109/L;
15. Patients with a platelet count ≤ 50.0x109/L;
16. Patients with aspartate aminotransferase (AST) or alanine aminotransferase (ALT) enzyme levels > 3 times the upper limit of normal during the 30 days prior to the transplant procedure;
17. Patients who were treated with any other investigational agent in the three months prior to enrolment;
18. Patients who received any investigational new drug, or participated in clinical study within the last 8 weeks;
19. Patient planned to receive an induction therapy different from rabbit ATG (Anti-thymocyte globulin) alone or patients who did not start rabbit ATG induction therapy after transplant;
20. Patients who are already on immunosuppressive drugs the day before transplantation, except ATG as per protocol;
21. Patients who are planned to receive therapy with any immunosuppressive agent other than those prescribed in the study;
22. Patients with a known hypersensitivity to corticosteroids, tacrolimus or everolimus or sirolimus or any of the excipients present in study drugs formulations;
23. Patients with hypersensitivity to macrolides;
24. Patients with any form of substance abuse, psychiatric disorder or a condition that, in the opinion of the Investigator, may invalidate communication with the Investigator;
25. Subjects unlikely to comply with the study protocol or unable to understand the nature and scope of the study but also the possible benefits or unwanted effects of the study treatments;
26. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-02-22 (Actual); Study Completion 2018-02-22 (Actual)

PRIMARY OUTCOMES:
Tacrolimus Area Under the curve at 24 hours (AUC24) | 10 days
Tacrolimus Minimum whole blood concentration (Cmin) | 10 days
Tacrolimus Cmin/daily dose | 10 days
Tacrolimus AUC24/daily dose | 10 days

SECONDARY OUTCOMES:
Tacrolimus within-patient variability of blood trough level | from day 3 to month 6
Time to reach therapeutic exposure to tacrolimus | from day 3 to month 6
Number of dose adjustments | from day 3 to month 6
Total daily dose | from day 3 to month 6
Renal function using estimated glomerular filtration rate | from day 1 to month 6
Treatment failure rate | from day 1 to month 6
Delayed graft function | from day 1 to month 6
  Number of days between the first and the last renal replacement session
Acute rejection requiring treatment | from day 1 to month 6
Biopsy proven acute rejections | from day 1 to month 6
Tacrolimus Maximum whole blood concentration (Cmax) | 10 days
Tacrolimus Tmax (time that the drug is present at the maximum concentration in serum) | 10 days
Tacrolimus Average whole blood drug concentration (Cave) | 10 days
Tacrolimus % fluctuation | 10 days
Tacrolimus % swing | 10 days
Tacrolimus linear correlation coefficient between Cmin and AUC24 | 10 days
Adverse Events | from screening to month 6
Serious Adverse Events | from screening to month 6
Number of opportunistic infections | from screening to month 6
  Number of opportunistic infections

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Rigotti, MD, Principal Investigator — Az Osp Padova, Osp. Civile Padova
Locations (6):
- Italy (6):
  - Ospedale Ca' Granda - Niguarda, Milan
  - Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera di Padova, Padua
  - Policlinico "A. Gemelli", Rome
  - Policlinico "Le Scotte", Siena
  - Azienda Ospedaliera S. Giovanni Battista, Torino

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/trial/2015-005640-34/results